CLINICAL TRIAL: NCT05930197
Title: An Exploratory Study of The Effect of Bismuth Subsalicylate on The Gut Microbiome and Host Response in Healthy Adults
Brief Title: Effect of Bismuth Subsalicylate on the Gut Microbiome and Host Response in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10001631; 001631-I
Record Dates: First submitted 2023-07-01; First posted 2023-07-05 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Healthy Adults
Keywords: Intestine; Gut; Metabolites; Microbiota
MeSH Terms: interventions — bismuth subsalicylate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): The oral suspension formulation of BSS will be used in this study. It is self administered at 1050mg 4 times per day (1 to 6 hours apart) for 2 days.
  Interventions: Drug: Bismuth subsalicylate

INTERVENTIONS:
Drug: Bismuth subsalicylate — BSS is a commonly used, widely available, OTC medication for a variety of gastrointestinal GI symptoms. It is available in the generic form, but also under the more commonly known brands: Bismatrol; Diotame; Geri-Pectate; Kao-Tin; Peptic Relief; Pepto-Bismol; Pink Bismuth and Stomach Relief. It received approval by the US Food and Drug Administration (FDA) in 1939.

SUMMARY:
Background:

Many kinds of good or normal bacteria live on your skin and inside your stomach and intestines (gut). These bacteria are important to your health. What you eat, where you live, and what medicines you take can affect the bacteria in your gut. Bismuth subsalicylate (BSS) is an ingredient in common medicines for mild diarrhea and stomach pain. Products that contain BSS include Pepto-Bismol, Kao-Tin, and Pink Bismuth. But how BSS affects the bacteria in a person s gut is not fully understood.

Objective:

To see how BSS affects gut bacteria in healthy people.

Eligibility:

Healthy people aged 18 to 50 years.

Design:

Participants will have 6 clinic visits in up to 18 weeks. Only 1 visit must be at the NIH clinic; others may be either in-person or remote.

BSS is a liquid taken by mouth. Participants will take a dose of BSS 4 times a day for 2 days. They will take the same amount of BSS as a person would take to treat diarrhea or related problems.

Stool samples will be collected at each study visit. For remote visits, participants will be given a collection kit; they will collect the sample at home and send it in.

Participants will take surveys at each visit. They will answer questions about their diet and health.

Participants may also provide optional samples of blood, saliva, and urine.

Participants may have up to 2 optional colonoscopies. A long tube will be inserted via the rectum to collect tissue samples from the intestine. Participants will be sedated or placed under anesthesia for the procedure.

DETAILED DESCRIPTION:
Study Description:

This is a single-site, single-arm, open-label study to evaluate the effect of bismuth subsalicylate (BSS) on the human gut microbiome and host immune response. Upon confirmation of eligibility, healthy adult volunteers will provide stool and optional blood, saliva, urine, and intestinal biopsy samples for a baseline assessment of gut microbiome and host immune response. Up to 18 weeks later, participants will undergo a 2-day/8-dose regimen of oral BSS. Stool will be collected at baseline, days 2 (+3), 8 (+/-3), 14 (-3/+7) and 28 (+/-7). Blood, saliva, and urine are also optional at these time points. Participants may also undergo a second optional colonoscopy at day 8 (+/-3) to provide colon biopsies for research analysis.

Primary Objective:

To evaluate the effect of BSS on the human gut microbiome.

Secondary Objective:

To evaluate the effect of BSS on the human gut metabolome.

Tertiary/Exploratory Objective:

To evaluate the effect of BSS on the systemic and intestinal host response (immune and inflammatory responses).

Primary Endpoint:

Differences in the relative abundance of taxa in stool samples pre-BSS and approximately 1 month post-BSS. Differences in microbiome metrics of alpha diversity and beta diversity will also be assessed.

Secondary Endpoint:

Differences in the stool metabolome (including short chain fatty acids, bile acids, and untargeted metabolomics) pre-BSS and approximately 1 month post-BSS.

Tertiary/Exploratory Endpoint:

Differences in systemic host immune and inflammatory responses, such as cytokines and immune cells, and host intestinal immune responses, such as specific T-cell populations in intestinal biopsies pre-BSS and approximately 1 month post-BSS.

ELIGIBILITY:
* INCLUSION CRITERIA:

An individual must meet all the following criteria to be eligible for this study:

* Aged 18 to 50 years.
* In generally good health.
* Able to provide informed consent.
* Willing to allow samples and data to be stored and shared for future research.
* Participants who can become pregnant must agree to use one effective method of contraception when engaging in sexual activities that can result in pregnancy, beginning at the signing of the informed consent form (as early as week -18) until the final study visit. Acceptable methods of contraception include the following:

  * External or internal condom with spermicide.
  * Diaphragm or cervical cap with a spermicide.
  * Hormonal contraception.
  * Intrauterine device.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Use of systemic antibiotics in the last 3 months.
* BSS use in the last 3 months.
* Pregnant or breastfeeding.
* Allergy to BSS.
* Allergy to other salicylates (including aspirin).
* Current use of other salicylates (including aspirin).
* Current use of anticoagulant medications.
* History of or active GI ulcers.
* History of or active bleeding disorder.
* Bloody stool within the last 3 months.
* Diarrhea within the last 2 weeks (defined as three or more loose or liquid stools per day).
* Current use of medications that may have a drug interaction with BSS.
* Not proficient in written English.
* Currently participating in another clinical trial that may affect current study procedures, per investigator s discretion.
* Any condition that, in the opinion of the study team, contraindicates participation in this study.

Co-enrollment in other studies is restricted. Consideration for co-enrollment in clinical trials evaluating the use of a licensed medication will require the approval of the principal investigator. Study staff should be notified of co-enrollment on any other protocol as it may require the approval of the principal investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Differences in the relative abundance of taxa in stool samples pre-BSS and approximately 1 month post-BSS. Differences in microbiome metrics of alpha diversity and beta diversity will also be assessed. | Through Day 28.
  To evaluate the effect of BSS on the human gut microbiome.

SECONDARY OUTCOMES:
Differences in the stool metabolome (including short chain fatty acids, bile acids, and untargeted metabolomics) pre-BSS and approximately 1 month post BSS. | Through Day 28
  To evaluate the effect of BSS on the human gut metabolome.

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra K Hourigan, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001631-I.html